CLINICAL TRIAL: NCT01594736
Title: Intracoronary Stenting and Angiographic Results: ORSIRO Stents Versus Xience PRIME Stents Assessed by Optical Coherence Tomography
Brief Title: ORSIRO Stents Versus Xience PRIME Stents Assessed by Optical Coherence Tomography
Acronym: ORSIRO_OCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MJ-MRI-ORSIRO_OCT-V3.1
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ORSIRO (Active Comparator)
  Interventions: Drug: ORSIRO
- XIENCE PRIME DES (Active Comparator)
  Interventions: Device: XIENCE PRIME DES

INTERVENTIONS:
Drug: ORSIRO — due randomization ORSIRO will be implanted
  Arms: ORSIRO
Device: XIENCE PRIME DES — due randomization XIENCE PRIME DES will be implanted
  Arms: XIENCE PRIME DES

SUMMARY:
This prospective, randomized trial will compare the extent of covered stent strut segments by assessed by Optical Coherence Tomography (OCT) of the ORSIRO DES with that of the XIENCE PRIME DES, which is the standard of choice of contemporary drug eluting stents (DES).

DETAILED DESCRIPTION:
The ORSIRO drug eluting stent exhibits a favourable vascular healing profile from baseline to 6 months assessed by optical coherence tomography (OCT). Patients with symptomatic coronary artery disease without cardiogenic shock who will undergo coronary angiography and willing to participate in the trial will receive before the procedure a loading dose of P2Y12 antagonists (clopidogrel, prasugrel or ticagrelor). Eligible patients who do not meet the exclusion criteria and for whom PCI will be considered as the appropriate form of revascularization will be randomly assigned to the ORSIRO or the XIENCE PRIME DES in the relation 1 x ORSIRO: 1 x XIENCE PRIME. All patients will receive periprocedural intravenous aspirin and heparin or bivalirudin. After the intervention patients will receive aspirin indefinitely and P2Y12 antagonists for at least 6 months. The intravascular imaging by OCT will be performed at the 6-8 months follow-up angiography.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than age 18 with ischemic symptoms or evidence of myocardial ischemia in the presence of ≥ 50% stenosis located in native coronary vessels.
* Written, informed consent by the patient or her/his legally-authorized representative for participation in the study.
* In women with childbearing potential a negative pregnancy test is mandatory.
* AHA type A, B1 and B2 lesions.

Exclusion Criteria:

* Lesion length > 25 mm requiring a stent length > 28 mm
* Target lesion located in the left main trunk.
* In-stent restenosis.
* Acute myocardial infarction
* Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than 18 months or that may result in protocol non-compliance.
* Known allergy to the study medications: sirolimus, everolimus
* Inability to take dual antiplatelet therapy for at least 6 months.
* The presence of bifurcation lesions
* The presence of calcified lesions
* Pregnancy (present, suspected or planned) or positive pregnancy test.
* Previous enrollment in this trial.
* Patient's inability to fully cooperate with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Degree of stent strut coverage at 6 months follow-up assessed by OCT for each visible strut segment | 6-18 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Joner, MD, Principal Investigator — Deutsches Herzzentrum München
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum München, Munich, Bavaria
  - Klinikum rechts der Isar, Munich, Bavaria